CLINICAL TRIAL: NCT02458573
Title: Comparison of the Effects of Continuous Epidural Analgesia and Continuous Intravenous Analgesia on Postoperative Bowel Movement in Patients Undergoing Laparoscopic Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2015-0157
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous epidural analgesia group (Experimental)
  Interventions: Other: continuous epidural analgesia
- continuous intravenous analgesia group (Active Comparator)
  Interventions: Other: continuous intravenous analgesia

INTERVENTIONS:
Other: continuous epidural analgesia — the continuous epidural analgesia group: epidural analgesia started from induction of anesthesia and continued for 48 h.
  Arms: continuous epidural analgesia group
Other: continuous intravenous analgesia — the continuous intravenous analgesia group: intravenous analgesia started from induction of anesthesia and continued for 48 h.
  Arms: continuous intravenous analgesia group

SUMMARY:
The investigators hypothesized that sympatholytic effect of epidural analgesia would attenuate the hemodynamic instability and decrease in the splanchnic blood flow caused by pneumoperitoneum during laparoscopic surgery. This study is to compare the effect of epidural analgesia and intravenous analgesia on postoperative bowel movement in patients undergoing laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 70 of age with ASA physical status Ⅰ-Ⅲ
* gastric cancer patient undergoing laparoscopic gastrectomy

Exclusion Criteria:

* ASA physical status Ⅳ
* bradycardia (< 60 bpm), arrhythmia
* uncompensated heart failure
* hepatic failure (Child-Pugh score B)
* renal failure (eGFR MDRD < 60 ml/min/1.73m2)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-03-28 (Actual)

PRIMARY OUTCOMES:
the time to first gas passing after surgery | within 5days after surgery
  Outcome will be assessed by a investigator blinded to the study group.
the time to resume water intake after surgery | within 5days after surgery
  Outcome will be assessed by a investigator blinded to the study group.
soft diet intake after surgery | within 5days after surgery
  Outcome will be assessed by a investigator blinded to the study group.

SECONDARY OUTCOMES:
postoperative pain | immediately after surgery to 48 hours
  numerical rating scale 0 (no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea